CLINICAL TRIAL: NCT05571267
Title: A Phase 2A Randomized Open-Label Controlled Trial to Assess the Safety of Zimura™ (Anti-C5 Aptamer) Administered in Combination With Anti-VEGF Therapy in Treatment Experienced Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Safety Study of Zimura in Combination With Anti-VEGF Therapy in Patients With Neovascular AMD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following Sponsor reassessment, OPH2004 enrollment was stopped to initiate a new Zimura wet AMD trial, OPH2007, for treatment-naïve patients. Thus, only one patient was enrolled into and completed Study OPH2004.
Sponsor: IVERIC bio, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPH2004
Record Dates: First submitted 2022-09-28; First posted 2022-10-07 (Actual); Results first posted 2023-04-03 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: Neovascular age-related macular degeneration (NVAMD)
MeSH Terms: interventions — Bevacizumab; Ranibizumab; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Avacincaptad Pegol and Avastin (Experimental): Participants receive three monthly Avastin treatments (Day 1, Month 1, and Month 2) followed by Avacincaptad Pegol administered on the same day. All participants will receive treatment every 3 months for a total of 18 months. If there is a loss of visual acuity during the intervening visits, participants may be retreated with Avastin and Avacincaptad Pegol.
  Interventions: Drug: Avacincaptad Pegol; Drug: Avastin
- Avacincaptad Pegol and Lucentis (Experimental): Participants receive three monthly Lucentis treatments (Day 1, Month 1, and Month 2) followed by Avacincaptad Pegol administered on the same day. All participants will receive treatment every 3 months for a total of 18 months. If there is a loss of visual acuity during the intervening visits, participants may be retreated with Lucentis and Avacincaptad Pegol.
  Interventions: Drug: Avacincaptad Pegol; Drug: Lucentis
- Avacincaptad Pegol and Eylea (Experimental): Participants receive three monthly Eylea treatments (Day 1, Month 1, and Month 2) followed by Avacincaptad Pegol administered on the same day. All participants will receive treatment every 3 months for a total of 18 months. If there is a loss of visual acuity during the intervening visits, participants may be retreated with Eylea and Avacincaptad Pegol.
  Interventions: Drug: Avacincaptad Pegol; Drug: Eylea

INTERVENTIONS:
Drug: Avacincaptad Pegol — Zimura 2 mg, administered by intravitreal injection
  Other Names: Zimura (previous name); IZERVAY; ARC1905
Drug: Avastin — Avastin 1.25 mg, administered by intravitreal injection
  Other Names: Bevacizumab
  Arms: Avacincaptad Pegol and Avastin
Drug: Lucentis — Lucentis 0.5 mg, administered by intravitreal injection
  Other Names: Ranibizumab
  Arms: Avacincaptad Pegol and Lucentis
Drug: Eylea — Eylea 2 mg, administered by intravitreal injection
  Other Names: Aflibercept
  Arms: Avacincaptad Pegol and Eylea

SUMMARY:
The primary objective is to assess the safety of intravitreal (IVT) Zimura® administered in combination with anti-VEGF Therapy (AVASTIN®, EYLEA®, OR LUCENTIS®) in anti-VEGF treatment experienced subjects with neovascular age-related macular degeneration (AMD)

ELIGIBILITY:
Inclusion Criteria:

* Treatment experienced subjects defined as subjects with 1 prior dose of same intravitreal anti-VEGF therapy given within the past 8 weeks for neovascular age-related macular degeneration (NVAMD) in the study eye. There must be < 0 letters of improvement in Snellen (not ETDRS Snellen equivalent) visual acuity since the start of anti-VEGF treatment.
* Presence of subfoveal active choroidal neovascularization (CNV)

Exclusion Criteria:

* Intravitreal treatment in the study eye prior to the Day 1 visit, regardless of indication, with the exception of the 1 prior anti-VEGF injections.
* Presence of other causes of choroidal neovascularization, including pathologic myopia, ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, and multifocal choroiditis.
* Non-pharmacologic treatment (intraocular surgery or thermal laser) within three months of trial entry.
* Prior thermal laser in the macular region, regardless of indication.
* Ocular or periocular infection in the past twelve weeks.
* History of any of the following conditions or procedures in the study eye: rhegmatogenous retinal detachment, pars plana vitrectomy, filtering surgery, glaucoma drainage device, or corneal transplant.
* Previous therapeutic radiation in the region of the study eye.
* Evidence of diabetic retinopathy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — IVERIC bio, Inc.

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=26399&tenant=MT_AST_9011
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/OPH2004/

RESULTS

PARTICIPANT FLOW:
Groups:
- Zimura and Avastin: Participants receive three monthly Avastin treatments (Day 1, Month 1, and Month 2) followed by Zimura administered on the same day. All participants will receive treatment every 3 months for a total of 18 months. If there is a loss of visual acuity during the intervening visits, participants may be retreated with Avastin and Zimura. Zimura: Zimura 2 mg, administered by intravitreal injection Avastin: Avastin 1.25 mg, administered by intravitreal injection
- Zimura and Lucentis: Participants receive three monthly Lucentis treatments (Day 1, Month 1, and Month 2) followed by Zimura administered on the same day. All participants will receive treatment every 3 months for a total of 18 months. If there is a loss of visual acuity during the intervening visits, participants may be retreated with Lucentis and Zimura. Zimura: Zimura 2 mg, administered by intravitreal injection Lucentis: Lucentis 0.5 mg, administered by intravitreal injection
- Zimura and Eylea: Participants receive three monthly Eylea treatments (Day 1, Month 1, and Month 2) followed by Zimura administered on the same day. All participants will receive treatment every 3 months for a total of 18 months. If there is a loss of visual acuity during the intervening visits, participants may be retreated with Eylea and Zimura. Zimura: Zimura 2 mg, administered by intravitreal injection Eylea: Eylea 2 mg, administered by intravitreal injection
Period: Overall Study
Arm/Group | Zimura and Avastin | Zimura and Lucentis | Zimura and Eylea
Started | 1 | 0 | 0
Completed | 1 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Following the Sponsor's reassessment of the Zimura development program, enrollment was stopped in this trial as the Sponsor determined that they would initiate a new Zimura wet AMD trial, the OPH2007 trial, for treatment-naïve patients. Therefore, a total of two patients were screened, one of whom was a screen failure. Thus, only one patient was enrolled into Study OPH2004.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zimura and Avastin | Zimura and Lucentis | Zimura and Eylea | Total
Number analyzed (Participants) | 1 | 0 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 0 | 0 | 1
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With >0 Letter Loss
Description: Vision testing is performed using retroilluminated modified Ferris-Bailey Early Treatment Diabetic Retinopathy Study (ETDRS) charts at 4 meters. Observed VA loss at Month 12 from Day 1 was assessed.
Time Frame: Month 12
Population: Only one patient was enrolled into Study OPH2004. This participant was included in the Zimura and Avastin arm. There were no participants in the Zimura and Lucentis arm and there were no participants in the Zimura and Eylea arm.
Measure: Number; unit: percentage of participants
Arm/Group | Zimura and Avastin | Zimura and Lucentis | Zimura and Eylea
Number analyzed (Participants) | 1 | 0 | 0
percentage of participants | 0 |  |

2. Primary Outcome: Percentage of Participants With >0 Letter Loss
Description: Vision testing is performed using retroilluminated modified Ferris-Bailey Early Treatment Diabetic Retinopathy Study (ETDRS) charts at 4 meters. Observed VA loss at Month 18 from Day 1 was assessed.
Time Frame: Month 18
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Zimura and Avastin | Zimura and Lucentis | Zimura and Eylea
Number analyzed (Participants) | 1 | 0 | 0
percentage of participants | 0 |  |

3. Primary Outcome: Percentage of Participants With >5 Letter Loss
Description: Vision testing is performed using retroilluminated modified Ferris-Bailey ETDRS charts at 4 meters. Observed VA loss at Month 12 from Day 1 was assessed.
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Zimura and Avastin | Zimura and Lucentis | Zimura and Eylea
Number analyzed (Participants) | 1 | 0 | 0
percentage of participants | 0 |  |

4. Primary Outcome: Percentage of Participants With >5 Letter Loss
Description: Vision testing is performed using retroilluminated modified Ferris-Bailey ETDRS charts at 4 meters. Observed VA loss at Month 18 from Day 1 was assessed.
Time Frame: Month 18
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Zimura and Avastin | Zimura and Lucentis | Zimura and Eylea
Number analyzed (Participants) | 1 | 0 | 0
percentage of participants | 0 |  |

5. Primary Outcome: Percentage of Participants With >10 Letter Loss
Description: as for outcome 3
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Zimura and Avastin | Zimura and Lucentis | Zimura and Eylea
Number analyzed (Participants) | 1 | 0 | 0
percentage of participants | 0 |  |

6. Primary Outcome: Percentage of Participants With >10 Letter Loss
Description: as for outcome 4
Time Frame: Month 18
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Zimura and Avastin | Zimura and Lucentis | Zimura and Eylea
Number analyzed (Participants) | 1 | 0 | 0
percentage of participants | 0 |  |

ADVERSE EVENTS:
Time Frame: Starting on Day 1, after first dose of trial drug, and continuing until 30 days after the last dose or until the last follow-up visit required by the protocol, whichever comes later, up to approximately 18 months.
Description: Only one patient was enrolled into Study OPH2004. This participant was included in the Zimura and Avastin treatment arm. There were no participants included in the Zimura and Lucentis arm and there were no participants included in the Zimura and Eylea arm.
Arm/Group | Zimura and Avastin | Zimura and Lucentis | Zimura and Eylea
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zimura and Avastin (N=1) | Zimura and Lucentis (N=0) | Zimura and Eylea (N=0)
nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Following the Sponsor's reassessment of the Zimura development program, enrollment was stopped in this trial as the Sponsor determined that they would initiate a new Zimura wet AMD trial, the OPH2007 trial, for treatment-naïve patients. Therefore, a total of two patients were screened, one of whom was a screen failure. Thus, only one patient was enrolled into Study OPH2004.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual site or investigator may publish or present any results from the trial until a joint, multi-center publication of the trial results is made by Sponsor in conjunction with various participating investigators and appropriate sites contributing data and comments. Subsequently, individual investigators may request to publish or present results from the trial; however approval will be at the sole discretion of the Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT05571267/Prot_SAP_000.pdf